CLINICAL TRIAL: NCT05088798
Title: Use of18F-DOPA PET/MRI for the Detection and Localization of Focal Forms of Hyperinsulinism
Brief Title: Utility of 18FDOPA PET/MRI for Focal Hyperinsulinism
Acronym: 18FDOPA HI
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Washington University School of Medicine (Other)
Collaborators: St. Louis Children's Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 201801029
Record Dates: First submitted 2021-06-18; First posted 2021-10-22 (Actual); Last update posted 2025-12-19 (Actual); Status verified 2025-12

CONDITIONS: Hyperinsulinism
Keywords: hypoglycemia; Glucose Metabolism Disorders; Infant, Newborn, Diseases; Hyperinsulinism; Insulinoma
MeSH Terms: conditions — Hyperinsulinism; Hypoglycemia; Glucose Metabolism Disorders; Infant, Newborn, Diseases; Insulinoma | interventions — fluorodopa F 18

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- 18F-Fluoro Dopa Imaging (Experimental): single arm
  Interventions: Drug: 18F-Fluoro Dopa PET/MRI Imaging

INTERVENTIONS:
Drug: 18F-Fluoro Dopa PET/MRI Imaging — The purpose of this research study is to provide access to an imaging study of the pancreas that uses 6-[18F]-Fluoro-L-3,4,-dihydroxyphenylalanine (18F-DOPA)positron emission tomography (PET) and assess the accuracy of this 18F-DOPA-PET/MRI test on distinguishing what part of the pancreas is affected in patients with Hyperinsulinism.
  Other Names: 6-[18F]-Fluoro-L-3,4,-dihydroxyphenylalanine; 18F-DOPA; [18F]-Fluorodopa

SUMMARY:
The purpose of the study is to provide access to 18F-DOPA PET to patients at Washington University and assess the utility of 18F-DOPA PET/MRI as a preoperative tool to detect and localize focal lesions in the pancreas that are causing hyperinsulinism.

DETAILED DESCRIPTION:
Congenital hyperinsulinism (CHI) is a clinically and genetically heterogeneous disorder that is the most common cause of permanent hypoglycemia in infants and children. More than 50% of the medically-unresponsive patients have focal disease. Which is characterized by a distinct region of Beta-cell hyperplasia in the pancreas, due to a somatic loss of a gene that regulates cell proliferation. Resection of the involved region cures most cases of focal HI. Therefore, preoperative identification and localization of focal HI lesions is useful for diagnostic confirmation and surgical guidance of patients with HI that fail pharmacological therapy and are being considered for surgery.

Insulinomas are benign insulin secreting neuroendocrine neoplasms located in the pancreas. They are the most common cause of endogenous hyperinsulinemic hypoglycemia in adults. Approximately 90% are solitary, benign and < 2cm in diameter and therefore represent a challenge to localize. The small size of insulinomas makes detection by conventional imaging techniques such as contrast-enhanced CT (ceCT) and contrast-enhanced MRI challenging. As surgery appears to be the only available treatment option, it remains very critical to localize the tumor to facilitate pancreas preserving surgery. Endoscopic ultrasound is well established in the detection of insulinomas. However, this technique is operator dependent, invasive, and the visualization of the pancreas tail is not always possible. Therefore better imaging techniques to detect these lesions are needed for surgical planning.

Though not FDA approved, noninvasive imaging with 18F-fluoro-L-DOPA (FDOPA) is considered an integral part of standards of care management to identify focal lesions in CHI and potentially insulinomas. This is based on the fact that 18F-DOPA is selectively taken up by neuroendocrine cells, and thus, in focal HI, dense collections of endocrine cells can be visualized by an experienced radiologist. This study aims to determine if using combined positron emission tomography and magnetic resonance imaging will better localize the lesions and help the investigators determine which areas of the pancreas are affected, and assist with the surgical plan.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with confirmed hyperinsulinemic hypoglycemia, diagnosed by elevated insulin levels during hypoglycemia and/or response to glucagon stimulation.
2. Subjects who failed pharmacological therapy with diazoxide or octreotide.
3. Subjects with signed informed consent by themselves or their parents or legal guardians.
4. Patient's Endocrinologist has determined that the patient cannot be safely managed with standard medical therapy (failed) and surgery is recommended to prevent future episodes of severe hypoglycemia and preserve brain function.

Exclusion Criteria:

1. Any other major illness or condition that in the investigator's judgment will substantially increase the risk associated with the subject's participation in this study.
2. Patient must not have any contraindication to MRI as evaluated by a standardized MRI safety questionnaire. If MRI is contraindicated, and patient meets inclusion criteria and has no other contraindications study will be conducted in PET/CT scanner.
3. Cases in which surgery will not be considered by parents or guardians.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2020-09-10 (Actual); Primary Completion 2030-01-01 (Estimated); Study Completion 2030-01-01 (Estimated)

PRIMARY OUTCOMES:
Increase Access to 18F-DOPA PET/MRI (or PET/CT) for patients with HI who failed medical therapy | one year
  To provide access to 18F-DOPA PET/MRI (or PET/CT) for patients with HI who do not respond to pharmacological therapy and are being considered for pancreatic surgery. We will measure this by totaling the number of scans performed yearly.

SECONDARY OUTCOMES:
Accuracy of 18FDOPA PET/MRI to identify focal forms of hyperinsulinism that may be cured by surgery | one year
  To identify if data from 18FDOPA PET/MRI imaging can accurately diagnose focal forms of HI when compared to the gold-standard of histopathological findings obtained at surgery in subjects who received a partial or complete pancreatectomy. Currently this type of isotope is not available for diagnosis, of insulinomas.

CONTACTS AND LOCATIONS:
Overall Officials: Ana Maria Arbelaez, MD, MSCI, Principal Investigator — Washington University School of Medicine
Locations (1):
- Washington University, St Louis, Missouri, United States

IPD SHARING:
Plan to Share IPD: Yes
We will share de-identified data with researchers at other institutions in a HIPPA compliant format.
Supporting Information: CSR
Time Frame: Data will be available upon request.
Access Criteria: PET Imaging data may be shared with other investigators in a HIPPA compliant manor for potential collaboration.